CLINICAL TRIAL: NCT04277559
Title: Comparison of the Effect of Patient Preferred Music on Postoperative Anxiety
Brief Title: The Effect of Music on Postoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, anesthesiology and reanimation specialist doctor, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: music
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-01

CONDITIONS: Anxiety Postoperative
Keywords: Patient preferential music; Postoperative anxiety; Classical music

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient preferential music (Active Comparator): The preference of the patients will be listened to preoperatively through the headphones.
  Interventions: Other: Patient preferential music
- Classical music (Active Comparator): Classical music (Four Seasons from Vivaldi) will be listened to preoperatively through the headphones.
  Interventions: Other: Classical music
- No music (Placebo Comparator): the patients will not listen.
  Interventions: Other: No music

INTERVENTIONS:
Other: Patient preferential music — Patients will listen to their preferred music through the headphones before surgery.
  Arms: Patient preferential music
Other: Classical music — Patients will listen to classical music through headphones before surgery.
  Arms: Classical music
Other: No music — Patients will not listen to music.
  Arms: No music

SUMMARY:
In this study, it is planned to compare the effect of listening to the music preferred by the patient and classical music on postoperative anxiety.

DETAILED DESCRIPTION:
Preoperative anxiety can be detected via structured and standardized screening by the State-Trait Anxiety Inventory (STAI) I and II. 225 patients scheduled for inguinal hernia surgery for any reason in the age range of 18-70 will be included in our study. Preoperative STAI I and II score (anxiety questionnaire) will be applied to each patient. The patients will be divided into three groups as preoperative patient preferential music, classical music and not played. The patient favorite music track and singer without limiting the kind of music or classical music will be played through the headphones. The STAI will be repeated at postoperative, the Numeric Rating Scale (NRS) and patient satisfaction will be measured at postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Undergo inguinal hernia surgery under general anesthesia,
* Being the ability to speak, read and write the Turkish language

Exclusion Criteria:

* Poor vision
* Significant hearing loss
* Dementia
* Active opioid use
* Regular use of anxiolytics or discontinuation of them on the day of surgery
* Unwillingness to participate in the study
* Unwillingness to listening to music

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Spielberg State-Trait Anxiety Inventory (STAI) score | 4 hours
  The test scores between 20 and 80, with higher scores indicating more generalized and stronger anxiety. Preoperative and postoperative STAI I score questions will be asked.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.
The quality of postoperative functional recovery (QoR-40) score | 24 hours
  The quality of postoperative functional recovery will assess using the QoR-40, which assesses physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item is rated on a 5-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score ranges from 40 (poorest quality of recovery) to 200 (the best quality of recovery). The QoR-40 will administer one day before surgery in outpatient clinics of anesthesiology, and before discharge from hospital on the first postoperative day.
Patient satisfaction score | 24 hours
  Patient satisfaction will assess prior to discharge using a Likert scale type (range, 1 to 7) verbally administered questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dışkapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Gölbaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akelma FK, Altinsoy S, Nalbant B, Ozkan D, Ergil J. Comparison of classical and patient-preferred music on anxiety and recovery after inguinal hernia repair: a prospective randomized controlled study. Perioper Med (Lond). 2024 Aug 14;13(1):89. doi: 10.1186/s13741-024-00434-3. PMID 39143577